CLINICAL TRIAL: NCT04880967
Title: Feasibility of an App to Measure Patient Stressors During Treatment in an Intensive Care Unit (ICU Feel Better App)- a Before-and-after Study
Brief Title: Feasibility of an App to Measure Patient Stressors in an Intensive Care Unit (ICU Feel Better App)- a Before-and-after Study
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: ICU Feel Better App
Record Dates: First submitted 2021-04-22; First posted 2021-05-11 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Group: Cohort of n=20 intensive care unit patients from the ages of 18 years will be collected.
  Participants of this cohort will not use the ICU Feel Better App.
- Experimental Group: Cohort of n=20 intensive care unit patients from the ages of 18 years will be collected. Participants of this cohort will have the opportunity to use the ICU Feel Better App every day from the second day after admission to the ICU until the day of discharge from ICU.

SUMMARY:
This study examines the feasibility and efficacy of a mobile application (app), which enables critically ill patients to report perceived patient stressors to their caregivers.

DETAILED DESCRIPTION:
For many critically ill patients, treatment in an intensive care unit (ICU) is very stressful, and for some of the patients it is a traumatic experience. The domains of patient stressors encompass physical stressors, mental health stressors, communication stressors, and environmental stressors. The experience of stressors during ICU is associated with a higher risk of worse outcomes including delirium, delayed recovery, and post-intensive care syndrome (PICS). In the context of inpatient intensive care medicine, health care professionals (HCP) have problems to correctly rate the extent of their patients' stress.

In this study, we examine the feasibility and efficacy of a stressor-reporting system based on a mobile application (app), which allows critically ill patients to evaluate by themselves the intensity of their stressors, and thus, to communicate their stress experience to HCPs.

In the first assessment phase of this study, outcome data of a cohort of n=20 patients will be collected (cohort A). Participants of cohort A will not use the ICU Feel Better App. In the second phase, outcome data of another n=20 patients (cohort B) will be collected. Participants of cohort B will have the opportunity to use the ICU Feel Better App from the second day after admission to the ICU until the day of discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in an ICU
* Duration of treatment ≥48h
* Age: 18 years and older
* Male, female, or divers gender

Exclusion Criteria:

* Poor language skills
* Statement in patient letter or living will that excludes participation
* Participation in another prospective treatment study with indication delirium
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in an ICU, aged 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Patient reported perceived severity of patient stressors | Time until discharge from the intensive care unit, an expected average of 10 days
  Patient reported perceived severity of patient stressors (Mean score of patient stressor list ). Range: 0-4, higher scores indicate higher stress. At day 2 or 3 of ICU treatment (before first use of the app) (t1), and at the day before or the day of discharge from ICU (t2).

SECONDARY OUTCOMES:
Mental distress | Time until discharge from the intensive care unit, an expected average of 10 days
  Mental distress is measured by Patient Health Questionnaire 4 [PHQ-4, range: 0-12, higher scores indicate higher distress]
Acute perceived stress | Time until discharge from the intensive care unit, an expected average of 10 days
  Acute perceived stress is measured by Stress Thermometer (range: 0-10, higher scores indicate higher stress)
State anxiety | Time until discharge from the intensive care unit, an expected average of 10 days
  State anxiety is measured with the Faces Anxiety Scale [FAS, range: 1-5, higher scores indicate higher anxiety]
Pain | Time until discharge from the intensive care unit, an expected average of 10 days
  Pain is measured with the Faces Pain Scale (range: 0-10, higher scores indicate higher pain)
Self-reported cognitive functioning | Time until discharge from the intensive care unit, an expected average of 10 days
  Self-reported cognitive functioning is measured with a list of problems of cognitive functions (range: 0-4, higher scores indicate worse cognitive functioning)
Incidence of delirium | Time until discharge from the intensive care unit, an expected average of 10 days
  Incidence of delirium is measured by CAM-ICU twice per day until
Length of stay | Time until discharge from hospital, an expected average of 20 days
  Length of stay is measured in days.
Length of intensive care unit stay | Time until discharge from the intensive care unit, an expected average of 10 days
  Length of intensive care unit stay is measured in days.
Duration of mechanical ventilation | Time until discharge from the intensive care unit, an expected average of 10 days
  Duration of mechanical ventilation is measured in hours.
APACHE II-Score | Time until discharge from the intensive care unit, an expected average of 10 days
  APACHE II score is measured by the Acute Physiology and Chronic Health Evaluation System II.
Medication | Time until discharge from the intensive care unit, an expected average of 10 days
  Medication is measured by data retrieved from the patient data management system.
Treatment | Time until discharge from the intensive care unit, an expected average of 10 days
  Treatment is measured by data retrieved from the patient data management system.
Diagnoses | Time until discharge from the intensive care unit, an expected average of 10 days
  Diagnoses are measured by ICD-10 codes retrieved from the patient data management system.
Mode of intensive care unit admission | Time until discharge from the intensive care unit, an expected average of 10 days
  Mode of intensive care unit admission is measured by admission data retrieved from the patient data management system.
Diagnosis of post-intensive care syndrome (PICS) | Up to one month
  Diagnosis of PICS is measured by an extensive clinical examination.
Log data per patient | Time until discharge from the intensive care unit, an expected average of 10 days
  Process data of app use: Log data per patient measured from start to end of app use
Stressor intensity- | Time until discharge from the intensive care unit, an expected average of 10 days
  Process data of app use: Stressor intensity measured from start to end of app use
Support of study personal | Time until discharge from the intensive care unit, an expected average of 10 days
  Number of app use trials with assistance of study personnel.
Acceptance of app | Time until discharge from the intensive care unit, an expected average of 10 days
  Patient reported acceptance of app use, daily until the end of app use
Usability of app | Time until discharge from the intensive care unit, an expected average of 10 days
  Patient reported usability of app, daily until the end of app use
Relevance and understandability of app stressor items | Time until discharge from the intensive care unit, an expected average of 10 days
  Patient reported relevance and understandability of app stressor items until the end of app use

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No